CLINICAL TRIAL: NCT03410680
Title: Evaluation of a Habit-formation and Gamification Intervention to Improve Adherence to Antiretroviral Therapy Among MSM Who Are New HIV Patients in Mexico
Brief Title: A Habit-formation and Gamification Intervention to Improve ART Adherence Among MSM HIV Patients in Mexico
Acronym: FUERTES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: Hospital Civil Juan I. Menchaca (Other); Hospital General de Occidente (Other); CAPASITS Villahermosa (Unknown)
Responsible Party: Principal Investigator, Sergio Bautista Arredondo, Director of Health Economics and Health Systems Innovations, Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1-233508
Record Dates: First submitted 2018-01-08; First posted 2018-01-25 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: HIV
Keywords: Antiretroviral Therapy; Adherence; HIV; Men who have sex with men; Sexual minorities; habit-formation; gamification
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Masking Description: The recruiting staff will not have access to the results of randomization prior to recruiting the participant.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Patients will receive the standard of care at the clinic. Questionnaires will be applied 4 times in a period of 10 months
- Intervention arm (Experimental): Each participant will receive FUERTES for a period of 4 months. It consists of receiving a habit-formation kit, which include an information and habit-formation tool that can be accessed through a web platform, a mobile app and a booklet; b) pill cases; c) a fidget cube; and f) a notebook. Patients will have the option of contacting a MD though WhatsApp regarding questions related to their treatment.
  After completing baseline a questionnaire, patients with a score of 2 for barriers that might affect their ART adherence will be assigned a coach. The coach will have 7 one-on-one sessions with the patient in a period of 4 months in order to catalyze ART adherence. MSM living with HIV who have been taking ART for >3 years will provide a one-time one-on-one peer support session
  Interventions: Behavioral: FUERTES

INTERVENTIONS:
Behavioral: FUERTES — The intervention focuses on antiretroviral therapy habit-formation among MSM living with HIV
  Other Names: STRONG
  Arms: Intervention arm

SUMMARY:
In general, several studies show that adherence to antiretroviral therapy (ART) among men who have sex with men (MSM) is low. Yet, high adherence to ART is essential-not only to improve the quality of life and survival rates among MSM living with HIV, but also to reduce HIV transmission among their partners. Our project aims to address this unmet need through a community-based habit-formation intervention, which incorporates elements of gamification. This intervention will provide MSM living with HIV who have been recently diagnosed and linked to care several tools to develop the habit of taking their medication and overcome disruptive adherence events (DAE) that would otherwise lead to treatment abandonment or lower adherence.

Between 2015 and 2017, the investigators conducted a study funded by CONACYT -the Mexican Council for Research-in two Mexican cities to involve MSM living with HIV in the design of an intervention to improve ART adherence. Results from this study show that at the beginning of ART, MSM living with HIV can benefit greatly from a habit-formation community-based intervention that includes support mechanisms to tackle the multiple barriers they face.

Using these findings, the investigators created FUERTES, an intervention with two main components: 1) the provision of a simple tool that MSM can access to learn how to develop an habit of taking their ART drugs, and 2) the support of a trained peer with background in psychology to help teach them how to overcome the myriad of barriers they may face in achieving medication adherence.

This is a multicentre, parallel, randomized, controlled trial. The project's aim is to pilot-test the intervention and document its implementation. Specifically, the investigators will assess the effect of the intervention on ART adherence among MSM living with HIV at four and ten months. Secondary outcomes include viral load and CD4 cell counts. They will also assess the scalability of the intervention by measuring the costs of the intervention. The duration of the project is two years starting December 2017. The researchers hypothesize that the FUERTES intervention will improve ART adherence among MSM living with HIV starting ART by at least 15%, measured by the medication possession ratio.

DETAILED DESCRIPTION:
FUERTES is an intervention with two main components: 1) the provision of a simple tool that MSM can access to learn how to develop an habit of taking their ART drugs, and 2) the support of a trained peer with background in psychology to help teach them how to overcome the myriad of barriers they may face in achieving medication adherence.

The first component includes providing each participant in the intervention arm with a habit-formation kit, which will include: 1) an information and habit-formation tool that can be accessed through a web platform, a mobile app and a booklet 2) a pocket pill-case; 3) a weekly pill organizer; 4) a water bottle containing a hidden pill case; 5) a fidget cube; and 6) a notebook and pen. Patients will also have access to a phone number to solve questions regarding HIV and ART with a medical doctor.

The second component includes providing social support to patients with high level of barriers that might influence the adherence to ART, through two mechanisms. Firstly, participants will receive professional psychologists will act as habit-formation coaches and will provide emotional support, sex education and referral to relevant health services. Secondly, they will receive one-on-one habit-formation support from MSM living with HIV who have been taking ART for several years, with the objective of reducing self-stigma and providing experience and reassurance that living a full and healthy life with HIV is possible.

ELIGIBILITY:
Inclusion criteria:

1. be MSM
2. be 18 or more years of age
3. treatment initiation between one day and one month ago, with expected continuation of treatment for the next ten months
4. literate Spanish
5. living in the metropolitan area of Guadalajara or Villahermosa
6. willing and able to provide written informed consent and contact information ( a phone number).

Exclusion criteria:

1. cisgender or transgender woman
2. transvestite, transgender or transsexual man
3. living with AIDS and taking four or more medicines for opportunistic infections
4. diagnosis of any neurologic, memory, sight or any other clinical illness that would prevent them answering the questionnaires
5. kidney disease with creatinine clearance below 50
6. presenting with acute liver failure or chronic liver failure
7. negative perception towards ART (ART as pharmaceutical lie, more harmful than beneficial)
8. the presence of a mental illness that requires a care assistant/guardian or treatment with psychiatric medication (e.g. schizophrenia, bipolar disorder, etc.)
9. participating in another research study to improve ART adherence
10. living on the street
11. unwilling to provide written informed consent or contact information

11) refusal to participate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Being a woman, a transgender man or transgender woman is an exclusion criteria for the study
Enrollment: 184 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in HIV viral load | Baseline (week 0), 1 month, 4 months, 10 months, 3 years
  Change from Baseline HIV viral load measured through medical chart abstraction (suppressed HIV viral load: ≤ 40 copies/mL).
Change in CD4 cell count | Baseline (week 0), 1 month, 4 months, 10 months, 3 years
  Change from Baseline CD4 cell count measured through medical chart abstraction.

SECONDARY OUTCOMES:
Change in ART adherence status | Baseline (1 month), 4 months, 10 months
  ART adherence will be assessed by different well-validated methods. In this study, ART adherence will be measured using medication possession ratio which measures participants' medication adherence using pharmacy refill information. We will also use a questionnaire based on the "AIDS Clinical Trials Group (ACTG) adherence follow up questionnaire", adapted after the pilot phase. We will administer this questionnaire through self-interview survey in a phablet. We will also use a 30 day recall question.
  While higher values indicate better levels of adherence, patients with adherence levels of 90% and above are regarded as ART-adherent while those with values less than 90% are not adherent to ART medications.
Change in antiretroviral therapy habit-strength | Baseline (1 month), 4 months, 10 months
  We will assess patient's habit strength using a self-report habit index questionnaire. We will administer this questionnaire through a self-interview survey in a phablet. We will average the scale scores. A high mean score will indicate greater habit strength.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Bautista-Arredondo, MSc, Principal Investigator — National Institute of public Health
Locations (3):
- Mexico (3):
  - Hospital Civil Nuevo Dr. Juan I. Menchaca, Guadalajara, Jalisco
  - Hospital General de Occidente, Guadalajara, Jalisco
  - CAPASITS Villahermosa, Villahermosa, Tabasco

IPD SHARING:
Plan to Share IPD: Yes
The data generated will be available publicly in 2020 in Dataverse, and it could be made available from the corresponding author upon reasonable request, for academic purposes.
Supporting Information: SAP
Time Frame: The data generated will be available publicly in Dataverse starting January 2020
Access Criteria: To be defined after data collection ends

REFERENCES:
- [Derived] Andrade-Romo Z, La Hera-Fuentes G, Ochoa-Sanchez LE, Chavira-Razo L, Aramburo-Muro T, Castro-Leon L, Amaya-Tapia G, Andrade-Perez JS, Bautista-Arredondo S. Effectiveness of an intervention to improve ART adherence among men who have sex with men living with HIV: a randomized controlled trial in three public HIV clinics in Mexico. AIDS Care. 2024 Jun;36(6):816-831. doi: 10.1080/09540121.2023.2299322. Epub 2024 Feb 29. PMID 38422450